CLINICAL TRIAL: NCT05774470
Title: Bradycardia Recognition and Detection in Young Infants Using the Owlet OSS 3.0 Monitor (Brady-I Study)
Brief Title: Bradycardia Recognition and Detection in Young Infants Part-I
Acronym: BRADY-I
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Owlet Baby Care, Inc. (Industry)
Responsible Party: Principal Investigator, Colm Travers, Assistant Professor of Pediatrics, University of Alabama at Birmingham
Other Study IDs: 300010237
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Neonatal Bradycardia; Hypoxemia of Newborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Owlet OSS 3.0 — The Owlet OSS 3.0 is a non-invasive monitoring device. The Sock secures the Sensor to the baby's foot. The Sensor measures the baby's SpO2, heart rate, and movement, and transmits the baby's readings to the Base Station. The Base Station records and monitors the baby's readings and can indicate prompts as needed based on the data sent from the Sensor.

SUMMARY:
This prospective cohort study will determine the diagnostic accuracy of the Owlet OSS 3.0 monitor for the detection of episodes of bradycardia and/or hypoxemia among infants.

DETAILED DESCRIPTION:
We will attach an Owlet monitor to infants for a 48-hour period. We will prospectively collect data from this device to determine the accuracy of bradycardia and hypoxemia detection compared with hospital monitors. In addition, we will collect simultaneous high-resolution real time cardiorespiratory data from Philips MP70 patient monitors at the University of Alabama at Birmingham.

ELIGIBILITY:
Inclusion Criteria:

* Off ventilatory support/NCPAP/HFNC and phototherapy for > 48 hours
* Less than one-year corrected age
* Current weight >1500 grams
* Parents/legal guardians have provided consent for enrollment

Exclusion Criteria:

* a major malformation
* a neuromuscular condition that affects respiration or causes apnea
* active skin breakdown or skin infection
* terminal illness or decision to withhold or limit support
* We will exclude data from infants who develop shock/sepsis or require ventilatory support or phototherapy during the study period.

Ages: 1 Day to 365 Days | Sex: All
Age Groups: Child
Study Population: Infants admitted to the neonatal intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-04-22 (Actual); Primary Completion 2023-07-29 (Actual); Study Completion 2023-07-29 (Actual)

PRIMARY OUTCOMES:
Bradycardia and/or hypoxemia | 48 hours
  The diagnostic accuracy of the Owlet OSS 3.0 monitor for detection of bradycardia <50/min and/or hypoxemia with SpO2 <80% episodes for ≥3 seconds during a 48-hour period.

SECONDARY OUTCOMES:
Bradycardia episodes | 48 hours
  The diagnostic accuracy of the Owlet OSS 3.0 monitor for episodes of bradycardia using alternative definitions of depth and duration (<50/min; < 80/min; < 100/min; lasting ≥ 10 seconds; lasting ≥ 20 seconds).
Hypoxemia episodes | 48 hours
  The diagnostic accuracy of episodes of intermittent hypoxemia of different severity and duration (<80%; <85%; lasting ≥ 10 seconds; lasting ≥ 20 seconds).
Diagnostic accuracy | 48 hours
  The false alarm rate and other key measures of diagnostic accuracy.
Limits of agreement | 48 hours
  The limits of agreement of overall heart rate and oxygen saturation recordings compared with hospital monitors.

CONTACTS AND LOCATIONS:
Overall Officials: Colm P Travers, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Hospital, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Travers CP, Nakhmani A, Armstead KM, Benz RL, Foshee KM, Carlo WA. Diagnostic accuracy of an over-the-counter infant pulse oximeter for cardiorespiratory events. Arch Dis Child Fetal Neonatal Ed. 2025 Dec 15;111(1):F13-F19. doi: 10.1136/archdischild-2025-328540. PMID 40355254